CLINICAL TRIAL: NCT02059226
Title: Evaluating an Internet-based Program for Anxious Youth: a Pilot RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mandi Newton (Other)
Collaborators: IWK Health Centre (Other)
Responsible Party: Sponsor-Investigator, Mandi Newton, Assistant Professor, University of Alberta
Organization: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00036087; CIHR (MOP119531) (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based CBT (Experimental): Internet-based cognitive behavioural therapy
  Interventions: Behavioral: cognitive behavioural therapy
- Internet-based resource page (Active Comparator): Static webpage
  Interventions: Other: Internet-based resource page

INTERVENTIONS:
Behavioral: cognitive behavioural therapy — Internet-based CBT
  Arms: Internet-based CBT
Other: Internet-based resource page — Static webpage
  Arms: Internet-based resource page

SUMMARY:
Anxiety is a common mental health problem for Canadian youth. Anxiety that is diagnosed as a disorder and serious enough to require treatment affects up to 10% of all youth by the age of 16. Anxiety disorders can have serious negative effects on a young person's personal relationships, school performance, and family life. These disorders may not be discovered by youth, parents and health care providers. Even if anxiety disorders are discovered, youth may not get the right therapy. Anxious youth can become sick if their anxiety is not treated properly.

The investigative team will carry out research to test Breathe, their new Internet-based treatment for youth with anxiety problems. Youth can use this treatment at home. Breathe includes information materials and personalized homework assignments to help anxious youth learn ways to manage anxiety.

This study is a pilot randomized controlled trial (RCT) with two groups, an Internet-delivered cognitive behavioural therapy (CBT) experimental group (Breathe) and a resource webpage (control group; considered treatment as usual for youth waiting for services). The investigators will evaluate several methodological processes and outcomes through the following objectives:

1. To evaluate the change in youths' anxiety (primary outcome) from pre- to post- intervention.
2. To estimate recruitment and retention rates for a full-scale RCT.
3. To estimate a sample size for a full-scale RCT.
4. To define the minimal clinically important difference (MCID) for the primary outcome measure.
5. To measure intervention acceptability.
6. To determine the use of co-interventions during the trial.
7. To conduct a preliminary economic analysis.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV social anxiety, generalized anxiety, anxiety not otherwise specified, or adjustment disorder as the primary clinical problem
* ability to read and write English
* regular access to a telephone and a computer system with high speed Internet service
* ability to use a computer to interact with web material
* youth aged 13-14 must have a consenting parent

Exclusion Criteria:

* youth with an anxiety problem that is not included above
* youth who receive cognitive behavioural therapy
* youth who cannot provide consent

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in anxiety at 8 weeks | at 8 weeks (i.e., post-intervention)
  Anxiety will be measured using the Multidimensional Anxiety Scale for Children (MASC2)

SECONDARY OUTCOMES:
Recruitment rate | at 27 months
Retention rate | at 30 months
Minimal Clinically Important Difference (MCID) | at 8 weeks (i.e., post-intervention)
  We will ask youth allocated to the intervention arm about a MCID. The MCID represents the minimum change considered meaningful from the youth's perspective such that they consider treatment worth participating in. We will use the MCID to determine intervention effectiveness in a full-scale trial. To estimate the MCID, we will use youths' global ratings of change on a 10-point Likert scale (-5 to +5), a commonly used anchor.
Intervention acceptability | at 8 weeks (i.e., post-intervention)
  Satisfaction will be measured to infer intervention acceptability, which will be measured in youth allocated to the treatment arm. A 10-item instrument will measure engagement and sense of privacy, expectations and usefulness, communication, and technical (intervention) management. For 10 statements, a 4-point Likert response format ranging from strongly agree to strongly disagree will be used. Scores will range from 10 to 40 with scores ≥ 30 indicating higher acceptability.
Co-intervention use | at 8 weeks (i.e., post-intervention)
  We will ask youth whether they used other health care resources during the study (e.g., emergency department visit, other treatments, medication) and reasons for this use (e.g., unmet need, medication prescribed before the study).
Resource use/costs | at 8 weeks
  The following will be reviewed: (i) software development and maintenance costs (for intervention maintenance and delivery), (ii) training and personnel costs for intervention, (iii) health care utilization data (e.g., self-reported visits to the emergency department, hospital admission), and (iv) other reported costs reported (i.e., time off from work/school).
Intervention adherence | at 8 weeks (i.e., post-intervention)
  Intervention adherence will also be measured to infer intervention acceptability. Intervention adherence will be measured by documenting the number of modules and homework tasks completed. We will also record the number of tailored modules completed by each youth (treatment arm) and site visits (control arm). These data will be collected through the intervention's software system.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Newton, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - University of Alberta; Alberta Health Services, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario

REFERENCES:
- [Derived] O'Connor K, Bagnell A, McGrath P, Wozney L, Radomski A, Rosychuk RJ, Curtis S, Jabbour M, Fitzpatrick E, Johnson DW, Ohinmaa A, Joyce A, Newton A. An Internet-Based Cognitive Behavioral Program for Adolescents With Anxiety: Pilot Randomized Controlled Trial. JMIR Ment Health. 2020 Jul 24;7(7):e13356. doi: 10.2196/13356. PMID 32706720
- [Derived] Newton AS, Wozney L, Bagnell A, Fitzpatrick E, Curtis S, Jabbour M, Johnson D, Rosychuk RJ, Young M, Ohinmaa A, Joyce A, McGrath P. Increasing Access to Mental Health Care With Breathe, an Internet-Based Program for Anxious Adolescents: Study Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2016 Jan 29;5(1):e18. doi: 10.2196/resprot.4428. PMID 26825111